CLINICAL TRIAL: NCT03311646
Title: Impact of Exclusive Use of Low Nicotine Cigarettes on Compensatory Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tracy Smith, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 950; R03DA045197 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-17 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: All participants experienced an NNC phase (baseline) and a VLNC phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotine Content Manipulation (Experimental): All participants receive normal nicotine content (NNC) cigarettes during Baseline and all participants receive very low nicotine content (VLNC) cigarettes during the very low nicotine content condition.
  Interventions: Other: Normal nicotine content cigarettes (NNC, Baseline); Other: Very low nicotine content (VLNC)

INTERVENTIONS:
Other: Normal nicotine content cigarettes (NNC, Baseline) — Participants will exclusively smoke research cigarettes that have a normal nicotine content for five days/four nights while staying in a hotel.
Other: Very low nicotine content (VLNC) — Participants will exclusively smoke research cigarettes that have a very low nicotine content for five days/four nights while staying in a hotel.

SUMMARY:
Smoking is the leading cause of preventable death in the United States. An FDA-mandated reduction in the nicotine content of cigarettes might reduce the health burden of tobacco by reducing the prevalence of smoking. The proposed project will test the impact of nicotine reduction on smoking behavior and smoke exposure in a setting where participants are restricted from using their usual brand cigarettes.

DETAILED DESCRIPTION:
Smoking is the leading cause of preventable death in the United States. An FDA-mandated reduction in the nicotine content of cigarettes might reduce the health burden of tobacco by reducing the prevalence of smoking. The proposed project will test the impact of nicotine reduction on smoking behavior and smoke exposure in a setting where participants are restricted from using their usual brand cigarettes.Smokers will be confined to a hotel for two hotel stays (five days/ four nights each) during which they will only have access to the investigational cigarettes provided to them. The nicotine content of the investigational cigarettes may differ between the two weeks. Participants will enter the hotel in groups of 10 and everyone in a given stay will receive the same investigational cigarette. The first aim will assess measures of smoke and nicotine exposure including urinary cotinine and expired carbon monoxide. The second aim will assess behavioral measures of smoking including cigarettes smoked per day and puff topography.

ELIGIBILITY:
Inclusion Criteria:

* male or female participants who are least 18 years old and smoke daily
* willing to stay in a hotel for two four-night stays during the prearranged dates

Exclusion Criteria:

* unwilling to use research cigarettes as part of the trial
* pregnant, trying to become pregnant, or breastfeeding
* additional smoking and health criteria determined at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Smith, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith TT, Koopmeiners JS, White CM, Denlinger-Apte RL, Pacek LR, De Jesus VR, Wang L, Watson C, Blount BC, Hatsukami DK, Benowitz NL, Donny EC, Carpenter MJ. The Impact of Exclusive Use of Very Low Nicotine Cigarettes on Compensatory Smoking: An Inpatient Crossover Clinical Trial. Cancer Epidemiol Biomarkers Prev. 2020 Apr;29(4):880-886. doi: 10.1158/1055-9965.EPI-19-0963. Epub 2020 Feb 26. PMID 32102910

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened for eligibility prior to the baseline condition. Participants were then required to return to the lab on a designated date to complete an additional drug screen and begin the hotel phase. Participants could withdraw or be lost to follow up between screening and baseline.
Groups:
- Very Low Nicotine Content: All participants receive normal nicotine content (NNC) cigarettes during baseline and all participants receive very low nicotine content (VLNC) cigarettes during the very low nicotine content condition.
Period: Overall Study
Arm/Group | Very Low Nicotine Content
Started | 31 (Number who were eligible and consented.)
Completed | 16 (Completed VLNC Condition)
Not Completed | 15
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 5
Not completed — PI Withdrawal for Positive Drug Screen | 4

BASELINE CHARACTERISTICS:
Population: This is not an intent to treat trial. Baseline characteristics are reported only for those participants who were included in the final (analyzed) sample.
Groups:
- Nicotine Content Manipulation: All participants receive normal nicotine content (NNC) cigarettes during Baseline and all participants receive very low nicotine content (VLNC) cigarettes during the very low nicotine content condition. During both the NNC and VLNC conditions, participants stay in a hotel and exclusively use the cigarettes provided to them. Each condition lasts four nights / five days. Baseline outcomes for the NNC condition are reported below, and VLNC condition outcomes are reported in the results section.
Arm/Group | Nicotine Content Manipulation
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 38.87 [26 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16
Education: Some College or More [Count of Participants; unit: Participants] | 8
Usual cigarette brand is menthol [Count of Participants; unit: Participants] | 7
Self-reported cigarettes per day at screening [Mean (Full Range); unit: cigarettes per day] | 14.75 [7 to 30]
Breath Sample (Expired Carbon Monoxide) [Mean (Standard Deviation); unit: parts per million] — Measure of short term smoke exposure, higher readings indicate more smoke exposure, While in the hotel, participants provided breath samples at 8am, 12pm, 4pm, 8pm beginning with 4pm on Day 1 and ending with 12pm on Day 5. Data from the NNC (baseline) condition are reported here.
  parts per million
    Day 1 (4pm) | 17.16 (6.95)
    Day 1 (8pm) | 31.26 (15.26)
    Day 2 (8am) | 23.97 (12.15)
    Day 2 (12pm) | 32.16 (16.32)
    Day 2 (4pm) | 32.78 (16.87)
    Day 2 (8pm) | 32.74 (16.87)
    Day 3 (8am) | 24.60 (10.16)
    Day 3 (12pm) | 30.30 (16.31)
    Day 3 (4pm) | 29.06 (16.83)
    Day 3 (8pm) | 30.72 (15.61)
    Day 4 (8am) | 21.94 (11.74)
    Day 4 (12pm) | 30.38 (16.74)
    Day 4 (4pm) | 31.61 (18.16)
    Day 4 (8pm) | 32.09 (17.65)
    Day 5 (8am) | 26.39 (14.19)
    Day 5 (12pm) | 33.95 (17.11)
Average cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes per day] — Average number of cigarettes smoked per day during the hotel phase. Participants collected cigarette butts and returned them at 12pm each day creating four 24-samples during both the NNC (baseline) and VLNC conditions. Data from the NNC (Baseline) Condition are reported here.
  cigarettes per day
    1st 24-hr sample | 17.69 (8.26)
    2nd 24-hr sample | 19.13 (7.87)
    3rd 24-hr sample | 19.13 (9.01)
    4th 24-hr sample | 21.88 (9.13)
Minnesota Nicotine Withdrawal Scale [Mean (Standard Deviation); unit: units on a scale] — Minnesota Nicotine Withdrawal Scale, A measure of nicotine withdrawal. Presented here is the total score, which has a range of 0 to 60, with higher scores indicating more withdrawal. Participants complete a self-report questionnaire on Days 2-5 during the hotel phase of the NNC (baseline) and VLNC conditions. Data from the NNC (Baseline) Condition are reported here.
  units on a scale
    Day 2 | 20.44 (4.46)
    Day 3 | 21.13 (5.02)
    Day 4 | 21.13 (4.47)
    Day 5 | 21.38 (4.56)
Questionnaire of Smoking Urges [Mean (Standard Deviation); unit: units on a scale] — Questionnaire of Smoking Urges, a Measure of craving, Presented here is Total Score, Range from 10-70, Higher scores indicate greater craving. Participants complete the Questionnaire of Smoking Urges on Days 2-5 of both the NNC (baseline) and the VLNC conditions. Data from the NNC (baseline) condition are not reported here.
  units on a scale
    Day 2 | 19.25 (10.50)
    Day 3 | 22.06 (12.13)
    Day 4 | 18.94 (12.91)
    Day 5 | 19.00 (10.58)

OUTCOME MEASURES:

1. Primary Outcome: Breath Sample (Expired Carbon Monoxide)
Description: Measure of short term smoke exposure, higher scores indicate more smoke exposure. While in the hotel, participants provided breath samples at 8am, 12pm, 4pm, 8pm beginning with 4pm on Day 1 and ending with 12pm on Day 5. Outcome here are from the VLNC condition. Baseline (NNC) data are reported in the baseline characteristics section.
Time Frame: 8am, 12pm, 4pm, 8pm beginning with 4pm on Day 1 and ending with 12pm on Day 5
Population: Results are presented for the 16 participants who completed both the NNC (baseline) and the VLNC conditions. Not an intent to treat trial.
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Very Low Nicotine Content
Number analyzed (Participants) | 16
parts per million
  Day 1 (4pm) | 18.77 (8.12)
  Day 1 (8pm) | 31.07 (18.74)
  Day 2 (8am) | 25.38 (14.51)
  Day 2 (12pm) | 30.49 (16.04)
  Day 2 (4pm) | 36.72 (24.68)
  Day 2 (8pm) | 35.66 (18.79)
  Day 3 (8am) | 26.06 (13.62)
  Day 3 (12pm) | 31.65 (18.59)
  Day 3 (4pm) | 31.90 (17.47)
  Day 3 (8pm) | 34.14 (17.81)
  Day 4 (8am) | 23.27 (14.28)
  Day 4 (12pm) | 24.82 (14.09)
  Day 4 (4pm) | 28.99 (16.03)
  Day 4 (8pm) | 30.03 (17.25)
  Day 5 (8am) | 22.22 (13.18)
  Day 5 (12pm) | 30.99 (17.07)
Statistical Analysis 1: Comparison: Very Low Nicotine Content; Comparison of carbon monoxide during VLNC condition to carbon monoxide during the NNC (baseline) condition; Test type: Other — A linear mixed-model was used. The model included terms for cigarette nicotine content (VLNC/NNC), time, cohort, a random effect for subject, and a nicotine content x time interaction. Interaction was dropped when nonsignificant. Reported below is the effect of nicotine content as well as the interaction p-value; p = 0.92, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-1.27 to 1.4] — Mean Difference = VLNC-NNC; Interaction p-value: p=0.27

2. Primary Outcome: Average Cigarettes Smoked Per Day
Description: Measure of smoking behavior. Participants returned smoked cigarette butts each day at 12pm, creating four 24-hr samples for each hotel phase (NNC and VLNC). Outcomes reported here are from the VLNC condition. Baseline (NNC) data are reported in the baseline characteristics section.
Time Frame: Participants returned smoked cigarette butts each day at 12pm, creating four 24-hr samples for each hotel phase. Data reported here are for the four 24-hr samples of the VLNC condition.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Groups:
- Very Low Nicotine Content: Participants will receive both normal nicotine content cigarettes and very low nicotine content cigarettes
  Normal nicotine content cigarettes: Participants will smoke research cigarettes that have a normal nicotine content
  Lower nicotine content cigarettes: Participants will smoke research cigarettes that have a lower nicotine content
Arm/Group | Very Low Nicotine Content
Number analyzed (Participants) | 16
Cigarettes per day
  1st 24-hr sample | 19.13 (11.99)
  2nd 24-hr sample | 22.38 (14.69)
  3rd 24-hr sample | 20.13 (13.11)
  4th 24-hr sample | 20.69 (13.31)
Statistical Analysis 1: Comparison: Very Low Nicotine Content; Comparison of cigarette per day during VLNC condition to cigarette per day during the NNC (baseline) condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.15, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = 1.13, 95% CI 2-sided [-0.41 to 2.66] — Mean Difference = VLNC-NNC; Interaction p=0.23

3. Secondary Outcome: Minnesota Nicotine Withdrawal Scale
Description: Measure of withdrawal, Total Score is presented here, Range from 0-60 with higher scores indicating greater withdrawal. Participants complete this self-report questionnaire on Days 2-5 during the NNC (Baseline) and VLNC conditions. Presented here are the scores from the VLNC condition. Data from the NNC (Baseline) conditions are reported in the baseline section.
Time Frame: Participants complete this self-report questionnaire on Days 2-5 during the NNC (Baseline) and VLNC conditions. Presented here are the scores from the VLNC condition.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Very Low Nicotine Content
Number analyzed (Participants) | 16
units on a scale
  Day 2 | 23.94 (8.39)
  Day 3 | 24.19 (7.02)
  Day 4 | 23.69 (7.51)
  Day 5 | 25.00 (9.36)
Statistical Analysis 1: Comparison: Very Low Nicotine Content; Comparison of Minnesota Nicotine Withdrawal Scale during VLNC condition to Minnesota Nicotine Withdrawal Scale during the NNC (baseline) condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 3.19, 95% CI 2-sided [1.77 to 4.60] — Mean Difference=VLNC-NNC; Interaction p=0.95

4. Secondary Outcome: Questionnaire of Smoking Urges
Description: Measure of craving, Range from 10-70, Higher scores indicate greater craving. Participants complete the Questionnaire of Smoking Urges on Days 2-5 of both the NNC (baseline) and VLNC Condition. Data here are from the VLNC Condition.
Time Frame: Participants complete the Questionnaire of Smoking Urges on Days 2-5 of both the NNC (baseline) and VLNC Condition. Data here are from the VLNC Condition.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Very Low Nicotine Content
Number analyzed (Participants) | 16
units on a scale
  Day 2 | 19.94 (10.95)
  Day 3 | 21.31 (14.47)
  Day 4 | 20.00 (14.32)
  Day 5 | 18.94 (11.86)
Statistical Analysis 1: Comparison: Very Low Nicotine Content; Comparison of carbon monoxide during VLNC condition to carbon monoxide during the NNC (baseline) condition; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.84, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-2.0 to 2.5] — Mean Difference = VLNC-NNC; Interaction p=0.94

ADVERSE EVENTS:
Time Frame: one month
Description: Adverse Events were recorded either when spontaneously reported at any time during the hotel phase or when participants answered yes to the following question "Have you had any negative changes in your physical or mental health since you've been in the hotel that you think might be related to study participation?" This question was asked on Day 5 of both the NNC (baseline) and VLNC conditions. Events reported below may have been reported during either condition.
Groups:
- Nicotine Content Manipulation: All participants receive normal nicotine content (NNC) cigarettes during Baseline and all participants receive very low nicotine content (VLNC) cigarettes during the very low nicotine content condition. During both the NNC and VLNC conditions, participants stay in a hotel and exclusively use the cigarettes provided to them. Each condition lasts four nights / five days. Adverse events reported below may have been reported during either the NNC or VLNC condition.
Arm/Group | Nicotine Content Manipulation
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 13/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Content Manipulation (N=16)
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3
Angry/Irritable/Frustrated Mood (General disorders) | 2
Heartburn (Gastrointestinal disorders) | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2
Headache (General disorders) | 2
Body Pain and Achiness (General disorders) | 2
Change in Appetite (Metabolism and nutrition disorders) | 1
Sleep Disturbances (General disorders) | 1
Craving to Smoke (General disorders) | 1
Bowel Movement Irregularity (Gastrointestinal disorders) | 1
Depressed Mood/ Sad (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Allergic Reaction (General disorders) | 1
Body Numbness (General disorders) | 1
Bug Bites (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT03311646/Prot_SAP_000.pdf